CLINICAL TRIAL: NCT01078571
Title: Safety and Effectiveness of Adalimumab (HUMIRA®) in Patients Diagnosed With Rheumatoid Arthritis (DALI Study)
Brief Title: Safety and Effectiveness of Adalimumab in Patients Diagnosed With Rheumatoid Arthritis
Acronym: DALI
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-077
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Results first posted 2011-10-25 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2011-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Biologic; Tumor Necrosis Factors blockers agents Monoclonal antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA patients in treatment with adalimumab (Humira): RA patients in treatment with adalimumab (Humira) at 40mg alternate weeks
  Interventions: Biological: adalimumab (HUMIRA®)

INTERVENTIONS:
Biological: adalimumab (HUMIRA®) — The primary objective of the study is to evaluate the safety and tolerability of adalimumab (HUMIRA®) treatment, administered both in monotherapy and combined therapy, in rheumatoid arthritis (RA) patients under usual practice conditions.
  Other Names: HUMIRA®; adalimumab

SUMMARY:
Adalimumab is one of the pharmacological treatments for rheumatoid arthritis (RA) of more recent marketing authorization, and as a result of this, there are only efficacy and safety data from clinical trials with controlled conditions.The study will evaluate the safety and effectiveness of adalimumab in the common clinical practice of RA treatment in Spain, with several types of patients showing concomitant treatments or diseases and compliance. Among the tumor necrosis factor antagonists safety studies, adalimumab safety has been the less investigated in the common clinical practice because of, as a result of its recent marketing, it was not included in the BIOBADASER (Data Base for Biological Products in Spain, Rheumatology Spanish Society), Biologic Products Database of the Spanish Society of Rheumatology ) in which was determined an association between infliximab therapy and the risk of developing active tuberculosis. To ensure the maintaining of the strict common physician practice (no prescription induction), and following the recommendations of the SER (Sociedad Española de Reumatología, Spanish Society of Rheumatology) consensus documents, it will be selected only those patients that were already in treatment with adalimumab (HUMIRA),(except patients involved in clinical studies with Adalimumab), and had shown good response, or those that fulfilled treatment indication in accordance with the SER recommendations and following the Summary of Products Characteristics of adalimumab (HUMIRA).

DETAILED DESCRIPTION:
Main objective

* To evaluate safety and tolerability of adalimumab (HUMIRA) treatment, administered both in monotherapy and combined therapy, in rheumatoid arthritis patients under usual practice conditions.

Secondary objectives

* To evaluate the effectiveness of the adalimumab (HUMIRA) treatment, administered both in monotherapy and combined therapy, in rheumatoid arthritis patients under usual practice conditions in accordance with SER recommendations:
* To evaluate the life quality associated to the adalimumab (HUMIRA) treatment, administered both in monotherapy and combined therapy, in rheumatoid arthritis patients under usual practice conditions.
* To describe the profile of patients who are in treatment with adalimumab (HUMIRA) biological therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients who underwent adalimumab treatment at least for the previous 4 months before baseline visit, who have a good therapeutic response to treatment and have not been involved in previous clinical studies with Adalimumab or
* Patients who previously to the baseline visit, have been prescribe adalimumab complying treatment indication according to SER (Sociedad Española de Reumatología, Spanish Society of Rheumatology) recommendations:
* Patients who had provided informed consent.
* Patients who have been prescribed adalimumab according to the Summary of Product Characteristics

Exclusion Criteria:

* Patients in whom a continued 12- months follow up is not anticipated.
* The contraindications specified in the Summary of Products Characteristics
* Hypersensibility to some of the components of the medication to administer.
* Any pathology shown by the patient that, according to medical criterion, contraindicates the treatment indicated in the protocol according to the Summary of Products Characteristics of adalimumab (HUMIRA®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatologist consultant
Sampling Method: Non-Probability Sample
Enrollment: 705 (Actual)
Dates: Start 2006-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Ruiz-Zorrilla, MD, Study Director — Abbott
Locations (40):
- Spain (40):
  - Site Reference ID/Investigator# 29714, A Coruña
  - Site Reference ID/Investigator# 29061, Algeciras
  - Site Reference ID/Investigator# 29710, Almería
  - Site Reference ID/Investigator# 29719, Barcelona
  - Site Reference ID/Investigator# 29054, Barcelona
  - Site Reference ID/Investigator# 29698, Barcelona
  - Site Reference ID/Investigator# 29063, Barcelona
  - Site Reference ID/Investigator# 29718, Barcelona
  - Site Reference ID/Investigator# 29720, Barcelona
  - Site Reference ID/Investigator# 29706, Cadiz
  - Site Reference ID/Investigator# 29052, Calella
  - Site Reference ID/Investigator# 29065, Cartagena
  - Site Reference ID/Investigator# 29713, Córdoba
  - Site Reference ID/Investigator# 29703, El Palmar
  - Site Reference ID/Investigator# 28607, Ferrol
  - Site Reference ID/Investigator# 5338, Girona
  - Site Reference ID/Investigator# 29701, Granada
  - Site Reference ID/Investigator# 29705, Huelva
  - Site Reference ID/Investigator# 29050, Ibiza Town
  - Site Reference ID/Investigator# 29708, Jaén
  - Site Reference ID/Investigator# 29709, Jerez de la Frontera
  - Site Reference ID/Investigator# 29711, L'Hospitalet de Llobregat
  - Site Reference ID/Investigator# 29716, Lugo
  - Site Reference ID/Investigator# 29038, Manacor
  - Site Reference ID/Investigator# 29712, Mataro, Barcelona
  - Site Reference ID/Investigator# 29700, Málaga
  - Site Reference ID/Investigator# 29051, Ourense
  - Site Reference ID/Investigator# 29699, Palma de Mallorca
  - Site Reference ID/Investigator# 29717, Pamplona
  - Site Reference ID/Investigator# 29704, Reus
  - Site Reference ID/Investigator# 29715, Santiago de Compostela
  - Site Reference ID/Investigator# 30823, Seville
  - Site Reference ID/Investigator# 29068, Seville
  - Site Reference ID/Investigator# 29064, Tarragona
  - Site Reference ID/Investigator# 29058, Valls
  - Site Reference ID/Investigator# 29055, Vic
  - Site Reference ID/Investigator# 29697, Vigo
  - Site Reference ID/Investigator# 29059, Vigo
  - Site Reference ID/Investigator# 29702, Vigo/Pontevedra
  - Site Reference ID/Investigator# 29053, Viladecans

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab Treatment: Participants with rheumatoid arthritis receiving treatment with adalimumab at 40 mg alternate weeks
Period: Overall Study
Arm/Group | Adalimumab Treatment
Started | 705
Safety Population | 675
Intent-to-treat (ITT) Population | 591
Completed | 590
Not Completed | 115
Not completed — Adverse Event | 36
Not completed — Lack of effectiveness | 36
Not completed — Reason not reported | 21
Not completed — Withdrawal by Subject | 12
Not completed — Lost to Follow-up | 8
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab (Humira)
Number analyzed (Participants) | 591
Age Continuous [Mean (Standard Deviation); unit: years] — Based on the ITT population minus 5 who did not report their age (586).
  years | 54.15 (12.43)
Sex/Gender, Customized [Number; unit: participants] — Based on the ITT population (591).
  participants
    Female | 461
    Male | 127
    Gender not reported | 3
Region of Enrollment [Number; unit: participants] — Based on the ITT population (591).
  participants
    Spain | 591
Time from Diagnosis of Rheumatoid Arthritis [Mean (Standard Deviation); unit: Years] — The number of years since the participant first received a diagnosis of rheumatoid arthritis. Based on the ITT population minus 91 who did not report the time since first diagnosis (500).
  Years | 8.56 (6.86)
Positivity of the Rheumatoid Factor [Number; unit: participants] — The number of participants testing positive or negative for rheumatoid factor. Based on the ITT population (591).
  participants
    Positive for Rheumatoid Factor | 460
    Negative for Rheumatoid Factor | 114
    Rheumatoid Factor Results Unknown or Missing | 17
Previous Rheumatoid Arthritis Treatment [Number; unit: participants] — Whether or not participants had taken medication for rheumatoid arthritis within the last 5 years. Based on the ITT population (591).
  participants
    Had previous rheumatoid arthritis treatment | 588
    No previous rheumatoid arthritis treatment | 3

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Adalimumab Treatment. Adverse Events: Medical Occurrence in a Patient or Clinical Investigation Subject Administered a Pharmaceutical Product and Which Does Not Necessarily Have a Causal Relationship With the Treatment
Description: The safety and tolerability of adalimumab was assessed at each study visit. The overall number of participants experiencing serious adverse events (SAEs), non-serious adverse events (AEs) and AEs that led to discontinuation are presented. The number of participants presenting with any serious or non-serious event at each particular study visit is also reported. Note that for the incidence data participants were counted multiple times if they experienced an adverse event at more than 1 visit. For additional information see Reported Adverse Events.
Time Frame: Baseline, 1, 4, 6, and 12 months
Population: This analysis was performed in the safety population of all participants who took at least 1 dose of adalimumab (675 participants).
Measure: Number; unit: Participants
Arm/Group | Adalimumab Treatment
Number analyzed (Participants) | 675
Participants
  Overall: Experienced a serious adverse event | 28
  Overall: Experienced a non-serious AE | 184
  Overall: Discontinued from study due to an AE | 36
  Incidence: At least 1 AE at Baseline | 53
  -- Incidence: At least 1 AE at 1 month | 49
  -- Incidence: At least 1 AE at 4 months | 50
  -- Incidence: At least 1 AE at 6 months | 47
  -- Incidence: At least 1 AE at 12 months | 51
  Incidence: At least 1 SAE at Baseline | 4
  -- Incidence: At least 1 SAE at 1 month | 4
  -- Incidence: At least 1 SAE at 4 months | 6
  -- Incidence: At least 1 SAE at 6 months | 6
  -- Incidence: At least 1 SAE at 12 months | 8

2. Secondary Outcome: Disease Activity Score (DAS 28) Index Mean Change From Baseline. The Disease Activity Score (DAS) is a Combined Index That Has Been Developed to Measure the Disease Activity in Patients With Rheumatoid Arthritis (RA).
Description: The DAS 28 index measures disease activity in rheumatoid arthritis and is derived from the number swollen/tender joints, laboratory tests of inflammation, and participant assessment of global health (by marking a 10 cm line from "very good" to "very bad"). Ranges were used to classify participants, with a higher score indicating worse control of disease: Remission (<= 2.6), Low Disease Activity (>2.6 to <=3.2), Moderate Disease Activity (>3.2 to <= 5.1) and High Disease Activity (>5.1). The mean change in DAS 28 score from baseline to final is presented.
Time Frame: Baseline and 12 months
Population: Mean change from baseline to 12 months included the ITT population of 310 de novo and 281 participants treated greater than 4 months.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Adalimumab (De Novo): Those participants to whom adalimumab had been prescribed for the first time 4 months or less before the baseline visit were classified as "de novo" participants.
- Adalimumab (Treated for Greater Than 4 Months): Participants who had been taking adalimumab for 4 months or longer.
Arm/Group | Adalimumab (De Novo) | Adalimumab (Treated for Greater Than 4 Months)
Number analyzed (Participants) | 310 | 281
Units on a scale | 1.62 (1.61) | 0.21 (1.23)

3. Secondary Outcome: Disease Activity Score (DAS 28) Index Percentage Change From Baseline. The Disease Activity Score (DAS) is a Combined Index That Has Been Developed to Measure the Disease Activity in Patients With Rheumatoid Arthritis (RA).
Description: The DAS 28 index measures disease activity in rheumatoid arthritis and is derived from the number swollen/tender joints, laboratory tests of inflammation, and participant assessment of global health (by marking a 10 cm line from "very good" to "very bad"). Ranges were used to classify participants, with a higher score indicating worse control of disease: Remission (<= 2.6), Low Disease Activity (>2.6 to <=3.2), Moderate Disease Activity (>3.2 to <= 5.1) and High Disease Activity (>5.1). The percentage reduction of baseline values is presented.
Time Frame: Baseline and 12 months
Population: Mean reduction from baseline to 12 months was calculated for the ITT population of 310 de novo and 279 participants treated greater than 4 months.
Measure: Mean (Standard Deviation); unit: Percentage reduction
Arm/Group | Adalimumab (De Novo) | Adalimumab (Treated for Greater Than 4 Months)
Number analyzed (Participants) | 310 | 279
Percentage reduction | 0.28 (0.34) | 0.01 (0.42)

4. Secondary Outcome: Clinical Evaluation of Rheumatoid Arthritis (RA). Clinical Evaluation in the Inclusion Visit and in Each One of the Study Visits.
Description: The treating physician was to clinically assess each participant at each study visit and report the number of painful and swollen joints. The mean number of painful or swollen joints for participants evaluated at each time point are presented by subgroup. The number of participants evaluated in each subgroup at each time point are also reported.
Time Frame: Baseline, 1, 4, 6, and 12 months
Population: This analysis was conducted in the ITT population of 591 participants who had assessments at each time point. The number of de novo participants and participants treated greater than 4 months who were analyzed at each time point are given in parentheses.
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Adalimumab (De Novo) | Adalimumab (Treated for Greater Than 4 Months)
Number analyzed (Participants) | 310 | 281
Joints
  Painful Joints at Baseline (n=310 and n =281) | 7.93 (6.31) | 2.22 (3.39)
  -- At 1 month (n=277 and n=203) | 4.11 (5.13) | 1.67 (3.07)
  -- At 4 months (n=292 and n=271) | 2.99 (4.14) | 1.76 (2.99)
  -- At 6 months (n=269 and n=267) | 2.53 (3.42) | 1.71 (2.86)
  -- At 12 months (n=255 and n=262) | 2.46 (3.33) | 1.61 (3.03)
  Swollen Joints at Baseline (n=310 and n=281) | 6.19 (5.01) | 1.39 (2.41)
  -- At 1 month (n=277 and n= 204) | 2.94 (3.89) | 1.03 (2.16)
  -- At 4 months (n=292 and n=272) | 2.33 (3.39) | 1.04 (2.10)
  -- At 6 months (n=269 and n=266) | 2.53 (3.42) | 1.00 (2.02)
  -- At 12 months (n=255 and n=262) | 1.73 (2.83) | 0.97 (2.00)

5. Secondary Outcome: Life Quality Assessment Health Assessment Questionnaire (HAQ Questionnaire) Mean Change From Baseline.
Description: Quality of life was assessed using the Health Assessment Questionnaire (HAQ). The HAQ is a self-reported scale used in studies of rheumatoid arthritis to assess areas such as dressing/grooming arising, eating, walking, reach, grip, maintaining hygiene, and daily activities. The global HAQ questionnaire was scored as follows: <1 = no/mild disability, 1 to 2 = moderate disability, and >2 = severe disability. An increased score indicates a worsening of the disability. The mean change in global HAQ score from baseline to 12 months is reported (baseline value - final value).
Time Frame: Baseline and 12 months
Population: The analysis was conducted for participants who had both baseline and 12-month global HAQ assessments.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Adalimumab (De Novo) | Adalimumab (Treated for Greater Than 4 Months)
Number analyzed (Participants) | 305 | 280
Units on a scale | 0.44 (0.67) | 0.05 (0.48)

6. Secondary Outcome: Life Quality Assessment Health Assessment Questionnaire (HAQ Questionnaire) Percentage Change From Baseline.
Description: Quality of life was assessed using the Health Assessment Questionnaire (HAQ). The HAQ is a self-reported scale used in studies of rheumatoid arthritis to assess areas such as dressing/grooming arising, eating, walking, reach, grip, maintaining hygiene, and daily activities. The global HAQ questionnaire was scored as follows: <1 = no/mild disability, 1 to 2 = moderate disability, and >2 = severe disability. An increased score indicates a worsening of the disability. The percentage change from baseline to 12 months (12-month score minus baseline score divided by baseline score) is presented.
Time Frame: Baseline and 12 Months
Population: The analysis was conducted for participants who had both baseline and 12-month global HAQ assessments.
Measure: Mean (Standard Deviation); unit: Percentage change
Groups:
- Adalimumab (Treatment for Greater Than 4 Months): Participants who had been taking adalimumab for 4 months or longer.
Arm/Group | Adalimumab (De Novo) | Adalimumab (Treatment for Greater Than 4 Months)
Number analyzed (Participants) | 297 | 238
Percentage change | 0.25 (0.79) | -0.09 (1.54)

7. Secondary Outcome: Radiological Evaluation of Rheumatoid Arthritis (RA).
Description: Treating physicians were asked to obtain a structural damage assessment by performing x-rays of the hands and feet approximately 1 year after the previous structural damage assessment that was done prior to the participant entering the study. The number of participants with radiological erosions evaluated at baseline and the 12-month visit are summarized by subgroup.
Time Frame: Baseline and 12 months
Population: This analysis was conducted in the intent-to-treat population (591 participants total).
Measure: Number; unit: Participant
Groups:
- Adalimumab (De Novo): Those participants to whom adalimumab had been prescribed for the first time four months or less before the baseline visit were classified as "de novo" participants.
- Adalimumab (Treated for Greater Than 4 Months: Participants who had been taking adalimumab for 4 months or longer.
Arm/Group | Adalimumab (De Novo) | Adalimumab (Treated for Greater Than 4 Months
Number analyzed (Participants) | 310 | 281
Participant
  Total number evaluated or not reported at Baseline | 310 | 281
  a) Radiological erosions present | 153 | 156
  b) Radiological erosions not present | 75 | 57
  c) Radiological erosions unknown | 54 | 50
  Total evaluated or not reported at 12 months | 310 | 281
  a) Radiological erosions present | 58 | 97
  b) Radiological erosions not present | 49 | 45
  c) Radiological erosions unknown | 135 | 97

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during the course of the study were reported in detail on case report forms. Adverse events occurring during the study were reported up to 30 days or 5 half-lives after the last dose of adalimumab.
Description: The safety population included all participants who received at least one dose of adalimumab (675 total). While 184 participants experienced a non-serious adverse event, 18 experienced non-serious adverse events that had an incidence greater than 1% and are presented in the Other Adverse Event table.
Arm/Group | Adalimumab Treatment
Serious Adverse Events (participants affected / at risk) | 28/675
Other Adverse Events (participants affected / at risk) | 18/675
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Treatment (N=675)
Acute coronary syndrome (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Pericarditis (Cardiac disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1
Abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 2
Bacteraemia/listeriosis (Infections and infestations) | 1
Diarrhoea/pyrexia/salmonellosis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Radius fracture/sternal fracture (Injury, poisoning and procedural complications) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab Treatment (N=675)
Respiratory tract infection (Infections and infestations) | 8
Urinary tract infection (Infections and infestations) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.